CLINICAL TRIAL: NCT02937974
Title: Evaluate the Efficacy of Xuebijing Injection in Acute Exacerbations of COPD：a Multicentre Randomised Controlled Trial
Brief Title: Evaluate the Efficacy of Xuebijing Injection in Acute Exacerbations of COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government); Navy General Hospital, Beijing (Other); Rocket Force General Hospital，Chinese People's Liberation Army (Unknown); 307 Hospital of PLA (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Lixin Xie, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WK-2016-HR-02; Chinese PLA General Hospital (Other: Chinese PLA General Hospital)
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Xuebijing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Xuebijing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xuebijing (Experimental): Xuebijing injection 50ml in 100ml of Normal Saline IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days
  Interventions: Drug: Xuebijing
- Placebo (Placebo Comparator): Normal Saline 150ml IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xuebijing — Xuebijing injection 50ml in 100ml of Normal Saline IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days
  Arms: Xuebijing
Drug: Placebo — Normal Saline 150ml IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days
  Arms: Placebo

SUMMARY:
Objective: A prospective multicenter randomized controlled trial to assess the efficacy and safety of Xuebijing injection for acute exacerbation of chronic obstructive pulmonary disease(AECOPD).

Methods: 254 AECOPD inpatients will be recruited in 6 hospitals in China over 2 years. They will be randomly assigned to Experimental group and Placebo group，Experimental: Xuebijing injection 50ml in 100ml of Normal Saline IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days；Placebo Comparator: Normal Saline 150ml IV, in 80mins, per 12 hours. administration of the agent for consecutive 5 days. Compare the following index between the two groups: Invasive mechanical ventilation rate, length of hospital stay, Treg cell,Th1,Th2,HLA-DR,CRP,PCT,IL-4,IL-6,IL-10,TNF-α，IFN-γ, APACHEⅡ, CAPS score.

DETAILED DESCRIPTION:
A prospective multicenter randomized controlled trial to assess the efficacy and safety of Xuebijing injection for acute exacerbation of chronic obstructive pulmonary disease(AECOPD).

ELIGIBILITY:
Inclusion Criteria:

1. Body weight≥40kg and ≤100kg
2. Diagnosis of COPD :(following Global initiative for Chronic Obstructive Lung Disease，GOLD2016)
3. Forced Expiratory Volume in 1 second of less than 70% predicted value after bronchodilator
4. Acute exacerbation of COPD: the clinical presentation of the patient complaining of an acute change of symptoms(baseline dyspnea,cough,and/or sputum production)that is beyond normal day-to-day variation.
5. Assessment of COPD Exacerbations: Medical History:severity of COPD based on degree of airflow limitation;Duration of worsening or new symptoms;Number of previous episodes (total/hospitalizations); Comorbidities; Present treatment regimen;Previous use of mechanical ventilation;
6. sign the informed consent

Exclusion Criteria:

1. Pregnant women, lactating women；
2. Be allergic to Xuebijing；
3. Acute exacerbation of COPD onset of more than 72 hours；
4. AECOPD with severe hypoxemia：oxygenation index <150 or received Endotracheal intubation invasive mechanical ventilation；
5. Participation in another experimental protocol within 30 days of study entry
6. Primary diseases：Asthma，Cystic fibrosis，Lung cancer，Tuberculosis，Pulmonary sarcoidosis，Pulmonary interstitial fibrosis，Malignant neoplasms，Blood system diseases，HIV；
7. Complications：Pulmonary embolism，shock，DIC，Unstable cardiovascular disease，Upper gastrointestinal bleeding，pneumothorax，Severe liver and kidney dysfunction；
8. Mental incompetence or active psychiatric illness
9. used the following drugs within 72 hours days of study entry：Ulinastatin，Tanreqing， Reduning，Qingkailing；
10. The investigator judged that the subject could not be completed or should not participate in the trial：Hemodialysis more than 1 mouth，Organ transplant patients with potential medical dispute.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Invasive mechanical ventilation rate | 28 days
  Invasive mechanical ventilation rate in %

SECONDARY OUTCOMES:
length of Hospital stay | 28 days
  Invasive mechanical ventilation rate in days

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, Professor, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Derived] Xie S, Yan P, Yao C, Yan X, Huo Y, Zhang J, Liu S, Feng Z, Shang H, Xie L. Efficacy and safety of Xuebijing injection and its influence on immunomodulation in acute exacerbations of chronic obstructive pulmonary disease: study protocol for a randomized controlled trial. Trials. 2019 Feb 18;20(1):136. doi: 10.1186/s13063-019-3204-z. PMID 30777117
- See also: 19729666 — https://www.ncbi.nlm.nih.gov/pubmed/?term=19729666